CLINICAL TRIAL: NCT01113489
Title: Assessment of Oxidative Stress Markers in the Upper and Lower Airways of Atopic Children Treated With Nebulized Beclomethasone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Mark Gjomarkaj, National Research Council, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0002565
Record Dates: First submitted 2010-04-15; First posted 2010-04-30 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-05

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- beclomethasone dipropionate suspension for nebulization (Experimental)
  Interventions: Drug: beclomethasone dipropionate
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: beclomethasone dipropionate — 400 mcg/1 ml b.i.d.
  Arms: beclomethasone dipropionate suspension for nebulization
Drug: placebo — 1 ml b.i.d.
  Arms: placebo

SUMMARY:
Although it is well known that the presence of uncontrolled inflammation in upper airways may compromise the control of asthma and may favor the progression of asthma toward more severe grades of disease, few studies addressed whether therapies aimed to control both upper and lower airway inflammation may be more effective in controlling asthma. Markers of oxidative stress and of inflammation such as Nitrotyrosine and IL-5 are increased in the airways of children with atopic asthma and correlated with the levels of oral and nasal FeNO, and with the grade of atopy. We hypothesize that the treatment with Beclometasone nebulized with a facial mask (for treating both upper and lower airways) will be able to reduce the production of oxidants as well as of IL5 in both districts thus promoting clinical and functional improvements in mild intermittent asthmatic children. The results provided by this study will contribute to further clarify the relationship between nasal and bronchial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* children with intermittent asthma and allergic rhinitis

Exclusion Criteria:

* children with acute respiratory symptoms in the last 4 weeks
* children with nasal polyposis or bronchial or respiratory tract infections
* children with a severe exacerbation of asthma resulting in hospitalization during the last month

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in level of oral and nasal fractional exhaled nitric oxide (FeNO) | Baseline, 4 weeks

SECONDARY OUTCOMES:
Change in peak expiratory flow (PEF) | Baseline, 4 weeks
change in visual analogue scale score for symptoms of rhinitis | Baseline, 4 weeks
change in obstructive sleep apnea syndrome score | Baseline, 4 weeks
change in forced vital capacity (FVC) | Baseline, 4 weeks
change in symptom scores of wheezing | Baseline, 4 weeks
change in forced expiratory volume in 1 second (FEV1) | Baseline, 4 weeks
change in level of IL-5 in exhaled breath condensate | Baseline, 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Immunopathology and Pharmacology of the Respiratory System Institute of Biomedicine and Molecular Immunology (IBIM) Italian National Research (CNR), Palermo, Italy